CLINICAL TRIAL: NCT00608673
Title: Pimecrolimus 1% Cream vs. Betamethasone Valerate 0.1% Cream in the Treatment of Facial Discoid Lupus Erythematosus: a Double-Blind Randomized, Pilot Study.
Brief Title: Comparing the Therapeutic Efficacy of Pimecrolimus Cream With Betamethasone Cream for Discoid Lupus Erythematosus
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shahid Beheshti University of Medical Sciences (Other)
Responsible Party: Behrooz Barikbin, M.D., Skin research centre, Shahid Beheshti University, M.C.
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 77
Record Dates: First submitted 2008-01-23; First posted 2008-02-06 (Estimated); Last update posted 2008-02-15 (Estimated); Status verified 2008-01

CONDITIONS: Discoid Lupus Erythematosus
Keywords: discoid lupus erythematosus; pimecrolimus 1% cream; betamethasone valerate 0.1% cream
MeSH Terms: conditions — Lupus Erythematosus, Discoid | interventions — pimecrolimus; Betamethasone Valerate

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Patients in arm one used twice daily pimecrolimus 1% cream on their facial discoid lupus erythematosus lesions for 8 weeks.
  Interventions: Drug: Pimecrolimus 1% cream
- 2 (Active Comparator): Twice daily betamethasone valerate 0.1% cream to facial lesions of discoid lupus erythematosus for 8 weeks
  Interventions: Drug: betamethasone valerate 0.1% cream

INTERVENTIONS:
Drug: Pimecrolimus 1% cream — a very thin coat of pimecrolimus 1% cream, twice daily topically to the facial lesions of discoid lupus erythematosus
  Other Names: Elidel
  Arms: 1
Drug: betamethasone valerate 0.1% cream — A very thin coat of betamethasone valerate 0.1% cream, twice daily to facial lesions of discoid lupus erythematosus for 8 weeks.
  Arms: 2

SUMMARY:
Discoid lupus erythematosus lesions are commonly treated with corticosteroids, but corticosteroids may induce side effects such as thinning of the skin or scarring. Therefore, an alternative medication with the same efficacy, but without the side-effects is sought after.

Pimecrolimus is a newer drug specially designed to treat inflammatory diseases of skin. Its efficacy in treating discoid lupus erythematosus has not been studied extensively yet. However studies performed till now show promising results. Long-term topical use of this medication has not shown any serious side-effects in other skin diseases.

In this study we aimed at comparing pimecrolimus efficacy with that of a common therapeutic choice, betamethasone valerate 0.1% cream, to see if pimecrolimus can be used as an alternative medication in treating discoid lupus erythematosus.

ELIGIBILITY:
Inclusion Criteria:

* Patients harboring discoid lupus erythematosus lesions on their face or neck

Exclusion Criteria:

* Patients with discoid lupus erythematosus in the setting of systemic lupus erythematosus
* Patients having a more disseminated disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-04; Primary Completion 2007-07 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Efficacy end points included a combined score based on evaluation of erythema, infiltration and squamation | 1st day, after 2, 4, 6 and 8 weeks of treatment

SECONDARY OUTCOMES:
Secondary outcome: Safety assessments included monitoring of adverse events | 1st day, after 2, 4, 6 and 8 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Behrooz Barikbin, M.D., Study Chair — Skin Research Center of Shahid Beheshti medical University
Locations (1):
- Shohada'e Tajrish Hospital, Tehran, Tehran Province, Iran